CLINICAL TRIAL: NCT04545047
Title: CSP #2030 - Observational Study of Convalescent Plasma for Treatment of Veterans With COVID-19
Brief Title: Observational Study of Convalescent Plasma for Treatment of Veterans With COVID-19
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2030
Record Dates: First submitted 2020-09-09; First posted 2020-09-10 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: COVID-19; Antibodies, viral/blood; adult; Human; Retrospective Studies; Immunization, Passive; Pandemics; Antibodies, Neutralizing; COVID-19 serotherapy; Severe acute respiratory syndrome coronavirus 2; Coronavirus Infections / therapy
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed: Veterans who received COVID-19 convalescent plasma therapy within 2 days of eligibility
  Interventions: Biological: COVID-19 convalescent plasma
- Unexposed: Veterans who did not receive COVID-19 convalescent plasma therapy

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — Convalescent plasma collected from individuals who have recovered from COVID-19
  Groups: Exposed

SUMMARY:
The purpose of this study is to assess whether convalescent plasma therapy is associated with reduced 30-day all-cause mortality in a population of Veteran inpatients with non-severe coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
The convalescent plasma (CP) of individuals who have recovered from COVID-19 may help reduce symptoms and mortality when given to ill patients infected with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Clinical trials are needed to provide definitive evidence of the benefits and harms of CP in the treatment of COVID-19. While clinical trials are underway, observational research plays a critical role in providing preliminary scientific evidence to guide clinical practice.

This observational study aims to estimate the association between CP therapy and mortality after 30 days in a sample of SARS-CoV-2-positive patients with non-severe illness. Patients include those hospitalized at a facility within the Veterans Health Administration (VHA) of the Department of Veterans Affairs (VA), the largest integrated healthcare system in the United States. Using VA electronic health record data, the study is designed to emulate a target trial of convalescent plasma transfusion and mortality. The primary exposure of interest is the use or non-use of COVID-19 convalescent plasma, and the primary outcome is 30-day all-cause mortality.

A nested trial design will be used, in which patients will be followed from each day in which eligibility criteria are met (while hospitalized and after date of first positive SARS-CoV-2 test) for 30 days. The association between CP therapy and mortality will be assessed using pooled logistic models to estimate 30-day cumulative incidence curves, risk differences, and hazard ratios. Inverse probability weighting derived from propensity scores will be employed to minimize confounding by indication and other biases.

ELIGIBILITY:
Inclusion Criteria:

* US Veterans aged 21-80 years old
* Hospitalized between May 1, 2020 and November 17, 2020 with a SARS-CoV-2 positive test, at a VA Medical Center where convalescent plasma had been administered to at least one patient and remained a current practice at that VA Medical Center
* SARS-CoV-2 positive test within 7 days before or after hospital admission
* Minimum oxygen saturation (measured within the past day) >=90%
* Vitals (pulse, respiration, temperature, systolic blood pressure) and acute labs (hemoglobin, platelet, white blood cells) measured within the past 2 days
* Albumin, Alanine Aminotransferase (ALT), creatinine measured within the past 30 days
* Weight measurement recorded in the past 2 years

Exclusion Criteria:

* Prior intubation, ventilation, high flow oxygen, extracorporeal membrane oxygenation (ECMO), dialysis, or vasopressors during current hospitalization
* Record of prior treatment with CP
* Received long-term care in a domiciliary or nursing home in the past 90 days
* First CP recipient at a site
* Less than 30 days of follow-up

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with non-severe COVID-19 who tested positive for SARS-CoV-2 infection during admission at a VA medical center or who were admitted as inpatients to a VA medical center within 30 days after a positive test for SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 5044 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L. Smith, PhD, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Michael J Gaziano, MD MPH, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data on SARS-CoV-2 testing, COVID-19 treatment, comorbidities, and other COVID-19-related information are available through the VA COVID-19 Shared Data Resource data domain within the VA Corporate Data Warehouse (CDW). Veterans Health Administration (VHA) researchers can request access to VHA data sources and data access tools for a research protocol approved by a VA Research and Development (R&D) Committee and reviewed by an Institutional Review Board (IRB). Information about requesting access to http://vaww.vhadataportal.med.va.gov/DataAccess/ResearchAcces (internal to VA).

REFERENCES:
- [Result] Cho K, Keithly SC, Kurgansky KE, Madenci AL, Gerlovin H, Marucci-Wellman H, Doubleday A, Thomas ER, Park Y, Ho YL, Sugimoto JD, Moore KP, Peterson AC, Hoag C, Gupta K, Jeans K, Klote M, Ramoni R, Huang GD, Casas JP, Gagnon DR, Hernan MA, Smith NL, Gaziano JM. Early Convalescent Plasma Therapy and Mortality Among US Veterans Hospitalized With Nonsevere COVID-19: An Observational Analysis Emulating a Target Trial. J Infect Dis. 2021 Sep 17;224(6):967-975. doi: 10.1093/infdis/jiab330. PMID 34153099
- See also: CSP #2030 Study Information — https://www.vacsp.research.va.gov/CSPEC/Studies/INVESTD-R/CSP-2030-convalescent-plasma-study.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study did not recruit patients but rather analyzed patients' VA electronic health record data. Eligibility was assessed through the examination of clinical and administrative data of US Veterans with non-severe COVID-19 who were hospitalized between1 May 2020 and 17 November 2020 at a VA medical center where convalescent plasma was a current practice.
Pre-assignment Details: We included patients in a trial on each day of eligibility (0, 1, 2) (person-trial). Each patient could be assigned to the plasma group once and to the non-plasma group up to 3 times. Because plasma patients could contribute non-plasma person-trials on eligible days prior to treatment, the sum of patients in the 2 groups (5,044) exceeds the number of eligible patients (4,755). Of 11,269 person-trials, there were 402 plasma trials (402 patients) and 10,867 non-plasma trials (4,642 patients).
Units Other Than Participants: person-trials
Groups:
- Exposed-Convalescent Plasma Group: Person-trials contributed by Veterans who received COVID-19 convalescent plasma therapy within 2 days of eligibility
  COVID-19 convalescent plasma: Convalescent plasma collected from individuals who have recovered from COVID-19
- Unexposed-Non-Plasma Group: Person-trials contributed by Veterans who did not receive COVID-19 convalescent plasma therapy
Period: Overall Study
Arm/Group | Exposed-Convalescent Plasma Group | Unexposed-Non-Plasma Group
Started | 402; 402 person-trials (402 unique patients assigned to 402 person-trials in Convalescent Plasma Group) | 4642; 10867 person-trials (4642 unique patients assigned to 10,867 person-trials in Non-plasma Group)
Completed | 402; 402 person-trials (402 unique patients assigned to 402 person-trials in Convalescent Plasma Group) | 4642; 10867 person-trials (4642 unique patients assigned to 10,867 person-trials in Non-plasma Group)
Not Completed | 0; 0 person-trials | 0; 0 person-trials

BASELINE CHARACTERISTICS:
Population: Because the study design allowed a patient enter a trial more than once, the sum of unique patients assigned to plasma and non-plasma groups (n=5,044) exceeds the number of eligible patients identified in the electronic health records (n=4,755).
Units Other Than Participants: Person-trials
Groups:
- Exposed-Convalescent Plasma Group: Veterans who received COVID-19 convalescent plasma therapy within 2 days of eligibility
  COVID-19 convalescent plasma: Convalescent plasma collected from individuals who have recovered from COVID-19
- Unexposed-Non-plasma Group: Veterans who did not receive COVID-19 convalescent plasma therapy
- Total: Total of all reporting groups
Arm/Group | Exposed-Convalescent Plasma Group | Unexposed-Non-plasma Group | Total
Number analyzed (Participants) | 402 | 4642 | 4755
Number analyzed (Person-trials) | 402 | 10867 | 11269
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (11.3) | 64.1 (12.0) | 64.2 (12.0)
Sex: Female, Male [Count of Units; unit: Person-trials]
  Female | 32 | 766 | 798
  Male | 370 | 10101 | 10471
Race/Ethnicity, Customized [Count of Units; unit: Person-trials]
  Race: White | 258 | 6194 | 6452
  Race: Black | 109 | 3814 | 3923
  Race: Other | 35 | 859 | 894
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.2 (7.1) | 31.0 (7.2) | 31.0 (7.2)
Smoking status [Count of Units; unit: Person-trials]
  Never | 109 | 2791 | 2900
  Current | 81 | 2836 | 2917
  Former | 74 | 1923 | 1997
  Unknown | 138 | 3317 | 3455
Cardiovascular disorder within past 5 years [Count of Units; unit: Person-trials] | 156 | 4663 | 4819
Chronic obstructive pulmonary disease [Count of Units; unit: Person-trials] | 119 | 2463 | 2582
Dementia [Count of Units; unit: Person-trials] | 29 | 816 | 845
Diabetes [Count of Units; unit: Person-trials] | 219 | 5145 | 5364
Hypertension [Count of Units; unit: Person-trials] | 307 | 7747 | 8054
Estimated glomerular filtration rate within past 30 days [Mean (Standard Deviation); unit: ML/min/1.73m2] | 75.3 (27.6) | 73.5 (27.8) | 73.5 (27.8)
In intensive care unit [Count of Units; unit: Person-trials] | 153 | 2204 | 2357
Glucocorticoid use [Count of Units; unit: Person-trials] | 215 | 2258 | 2473
Remdesivir use [Count of Units; unit: Person-trials] | 187 | 1476 | 1663
Supplemental non-high-flow oxygen [Count of Units; unit: Person-trials] | 9 | 161 | 170
Minimum oxygen saturation in past day [Mean (Standard Deviation); unit: Percentage of oxyhemoglobin saturation] | 93.3 (2.8) | 94.6 (3.1) | 94.5 (3.1)
First oxygen saturation during hospitalization [Mean (Standard Deviation); unit: Percentage of oxyhemoglobin saturation] | 93.8 (3.8) | 95.5 (3.3) | 95.4 (3.4)
Maximum white blood cell count in past 2 days [Mean (Standard Deviation); unit: 1000 cells/ul] | 7.4 (4.1) | 6.8 (3.9) | 6.8 (3.9)
Systemic inflammatory response syndrome [Count of Units; unit: Person-trials] | 243 | 4739 | 4982
Calendar day of trial start [Mean (Standard Deviation); unit: days] | 249 (52) | 231 (52) | 232 (52)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Death at 30 days recorded in the electronic health record. Follow-up starts at the treatment date, which must be within 2 days after both hospitalization and SARS-CoV-2-positive test, and ends at 30 days or death.
Time Frame: 30 days
Population: Intention-to-treat analysis; per-protocol analysis with adjustment for baseline covariates via inverse probability weighting
Measure: Count of Units; unit: Person-trials
Units Other Than Participants: Person-trials
Groups:
- Convalescent Plasma Group: Veterans who received COVID-19 convalescent plasma therapy within 2 days of eligibility
  COVID-19 convalescent plasma: Convalescent plasma collected from individuals who have recovered from COVID-19
- Non-plasma Group: Veterans who did not receive COVID-19 convalescent plasma therapy
Arm/Group | Convalescent Plasma Group | Non-plasma Group
Number analyzed (Participants) | 402 | 4642
Number analyzed (Person-trials) | 402 | 10867
Person-trials | 40 | 671
Statistical Analysis 1: Comparison: Convalescent Plasma Group vs Non-plasma Group; The investigators estimated the 30-day mortality risk difference comparing patients assigned to each group. Adjustment for covariates would be carried out via inverse probability weighting; Test type: Superiority; Risk Difference (RD) = 0.30, 95% CI 2-sided [-2.30 to 3.60]
Statistical Analysis 2: Comparison: Convalescent Plasma Group vs Non-plasma Group; The investigators estimated the 30-day mortality hazard ratio comparing patients assigned to each group. The hazard ratio was estimated from pooled logistic models with inverse probability weighting to adjust for confounding; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.64 to 1.62]

ADVERSE EVENTS:
Time Frame: 30 days
Description: No adverse event data were collected for this retrospective observational EHR-based study
Groups:
- Convalescent Plasma Group: Veterans who received COVID-19 convalescent plasma therapy within 2 days of eligibility
Arm/Group | Convalescent Plasma Group | Non-plasma Group
All-Cause Mortality (participants affected / at risk) | 40/402 | 343/4642
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04545047/Prot_SAP_000.pdf